CLINICAL TRIAL: NCT02152930
Title: The Effects of Fish Oil Supplements During Supervised Exercise Therapy in Patients With Intermittent Claudication
Acronym: FISHTIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, Alexander P.J. Houdijk, Dr., Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL46719.029.13
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Intermittent Claudication
Keywords: Fish oil supplements; Supervised Exercise Training; Walking distance; Hemorheological factors; Cardiovascular risk
MeSH Terms: conditions — Intermittent Claudication | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised Exercise Therapy (Active Comparator): Standard treatment: Supervised Exercise Therapy during 12 weeks
  Interventions: Drug: Omega-3 fatty acids
- Controlled group (No Intervention)

INTERVENTIONS:
Drug: Omega-3 fatty acids — 1000 mg of omega-3 fatty acid ethylesters, 2 times daily, for 4 weeks, followed by 12 weeks of supervised exercise therapy in combination with 2 times daily omega-3 fatty acid supplementation.
  Other Names: Fish oil supplements
  Arms: Supervised Exercise Therapy

SUMMARY:
Intermittent claudication (IC) is caused by peripheral arterial disease and has a high morbidity and mortality. Etiologic factors are similar to those of cardiovascular disease. Primary treatment consists of cardiovascular risk management and improvement of functional capacity with supervised exercise therapy (SET). A potential additional therapy is the administration of fish oil supplements containing high amounts of omega-3 Poly Unsaturated Fatty Acids (PUFAs). In earlier clinical and experimental trials omega-3 PUFA's improved hemorheological parameters such as erythrocyte deformability and aggregation, and a number of cardiovascular risk factors. Hemorheological parameters determine the blood flow in the microcirculation, which is of main importance in patients with IC since the macrocirculation is compromised. Inflammation is considered an important etiologic factor in the pathogenesis of atherosclerosis and contributes to peripheral arterial disease Since omega-3 PUFAs also have a strong anti-inflammatory effect, they might be effective in patients with IC by lowering the inflammatory response. In addition, visceral fat rather than obesity in general has been recognised as an etiologic and prognostic factor in atherosclerosis.

We hypothesise that the administration of omega-3 PUFA's in patients with IC has a synergistic effect with SET and improves walking distance after SET, by improving hemorheological parameters resulting in a better microcirculation. Second, we hypothesise that omega-3 PUFA's result in a less proinflammatory of whole blood in response to ex vivo stimulation with endotoxin. Third, we hypothesise that omega-3 PUFA's and SET result in a decrease in visceral fat mass.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Newly diagnosed intermittent claudication
* Ankle Brachial Index < 0.8 at rest or > 0.15 decrease after exercise
* Able to perform standardised treadmill walking test for 2 min
* Written informed consent

Exclusion Criteria:

* Unable to fill out a questionnaire (cognitive impairment or insufficient knowledge of the Dutch language)
* Heart failure or unstable cardiac status (angina pectoris class III or IV or recent myocardial infarction < 3 months)
* Any illness with rapid evolution or a life expectancy < 3 months
* Recent cerebrovascular accident (< 3 months)
* Current use of fish oil supplements or > 2 times a week dietary fish
* Pregnancy
* Fish, soybean or peanut allergy
* Contra indications for the use of omega-3 fatty acids
* Use of oral anticoagulants (coumarin derivatives)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximal walking distance with standardised treadmill test | After 12 weeks of supervised exercise therapy

SECONDARY OUTCOMES:
Hemorheological parameters | After 12 weeks of supervised exercise therapy
Visceral fat mass | After 12 weeks of supervised exercise therapy
Ex vivo cytokine production after stimulation with lipopolysaccharide | After 12 weeks of supervised exercise therapy
Assessment of the microcirculation with side stream dark field technology | After 12 weeks of supervised exercise therapy

OTHER OUTCOMES:
Bloodpressure, heart rate, cholesterol, triglycerides, hemoglobin, leucocytes, C-reactive protein, ankle brachial index, | After 12 weeks of supervised exercise therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P.J. Houdijk, Dr., Principal Investigator — Medical Center Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands